CLINICAL TRIAL: NCT05215613
Title: PMCF Study to Provide Safety, Performance and Clinical Benefits Data of the Zimmer® Plates and Screws System Applied for Diaphyseal, Proximal Humerus and Proximal Tibia Fractures (Implants and Instrumentation) - A Retro- and Prospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the Zimmer® Plates and Screws System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-158T
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-11

CONDITIONS: Proximal Humeral Fracture; Proximal Tibia Fractures; Diaphyseal Fracture
Keywords: Medical device; Performance; Safety; Clinical benefits; Diaphysis; Proximal humerus; Proximal Tibia; Fracture; Post Market Clinical Follow Up Study
MeSH Terms: conditions — Shoulder Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients implanted with the Zimmer® Plates and Screws System: Patients who already received the Zimmer® Plates and Screws System in the Diaphysis, Proximal Humerus and Proximal Tibia.

SUMMARY:
The study is a monocentric, retro- and prospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to confirm safety, performance and clinical benefits of the Zimmer® Plates and Screws System (implants and instrumentation) when used to stabilize diaphyseal, proximal humerus and proximal tibia fractures.

The primary objective is the assessment of performance by analyzing fracture healing.

The secondary objectives are the assessment of safety by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified. Subjects' outcomes will also be assessed.

DETAILED DESCRIPTION:
The Zimmer® Plates and Screws System consists of temporary internal fixation devices comprised of plates and screws that provide management of fractures through interfragmentary compression and bone plating. In this study, the focus is on the Zimmer® Plates and Screws System used to stabilize diaphyseal, proximal humerus and proximal tibia fractures.

One site will be involved in this study. The aim is to include a maximum of 112 consecutive series cases who received the Zimmer® Plates and Screws System at the Istituto Ortopedico Rizzoli (Bologna, Italy) between 2008 and 2018. All potential study subjects will be required to participate in the Informed Consent process.

Baseline data from the preoperative, intraoperative, immediate post-operative and last consultation visit at minimum 6 months post-operative will be available in medical notes and collected retrospectively. During a follow up phone call the subject will be asked to complete questionnaires and a clinical assessment of the fracture healing. In addition, any complications since the last consultation visit at the clinic and information about the treatment of the complications will also be collected over the phone.

ELIGIBILITY:
Inclusion Criteria:

Patients having received one of the plates belonging to the Zimmer® Plates and Screws System, designed for temporary internal fixation to stabilize fractures during the normal healing process. In this study we will collect data specifically on Zimmer® Plates and Screws System plates belonging to the Diaphysis, Proximal Humerus and Proximal Tibia groups.

Exclusion Criteria:

* Off-label use
* Patients under the age of 18
* Prisoners
* Severely comminuted fractures in which bone fragments are too small or numerous to adequately fix or maintain a reduced position
* Infection
* Metal sensitivity or intolerance
* Severe osteopenia and/or osteoporosis, or in the presence of marked or rapid bone absorption, metabolic bone disease, cancer, or any other tumor-like condition of the bone which may compromise fixation
* Sternal or spinal fractures
* Anatomical location in which the device would interfere with nerves, blood vessels, or other vital structures
* Patients with inadequate soft tissue coverage at the implant site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of cases implanted with plates and screws belonging to the Zimmer® Plates and Screws System according to Zimmer Biomet's Instruction for Use (IFU) and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- SC Clinica Ortopedica e Traumatologica II IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient's fracture was revised with the study device and was therefore enrolled twice as 2 separate cases in the study, as two study devices were used.
Units Other Than Participants: Fracture
Groups:
- Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate: 30 participants (31 cases) who meet the inclusion and none of the exclusion criteria and who received the Zimmer® Plates and Screws System in the Diaphysis.
- Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate: 26 participants (26 cases) who meet the inclusion and none of the exclusion criteria and who received the Zimmer® Plates and Screws System in the Proximal Tibia.
Period: Overall Study
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate
Started | 30; 31 Fracture | 26; 26 Fracture
Completed | 30; 31 Fracture | 26; 26 Fracture
Not Completed | 0; 0 Fracture | 0; 0 Fracture

BASELINE CHARACTERISTICS:
Units Other Than Participants: Fractures
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate | Total
Number analyzed (Participants) | 30 | 26 | 56
Number analyzed (Fractures) | 31 | 26 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (19.6) | 36.2 (13.6) | 38.2 (17.1)
Sex: Female, Male [Count of Units; unit: Fractures]
  Female | 9 | 10 | 19
  Male | 22 | 16 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Concomitant Diseases [Count of Units; unit: Fractures]
  None | 25 | 17 | 42
  Cardiac / Respiratory Disease and Hypertension | 2 | 1 | 3
  Vascular Disease and Hypertension | 1 | 1 | 2
  Congenital Hip Dysplasia | 0 | 2 | 2
  Vascular Disease and Venous Insufficiency Right Lower Limb | 0 | 1 | 1
  Hypothyroidism | 0 | 1 | 1
  Osteogenesis Imperfecta | 0 | 1 | 1
  Cardiac / Respiratory Disease, Hypertension and Hypercholesterolemia | 1 | 0 | 1
  Diabetes and Hypercholesterolemia | 1 | 0 | 1
  Cardiac / Respiratory Disease, Hypertension, Hypercholesterolemia and Diabetes | 1 | 0 | 1
  Prothrombin Gene Mutation | 0 | 1 | 1
  Previous Open Fracture and Internal Fixation Right Femur and Patella 1 year earlier | 0 | 1 | 1
Confounding fractures for bone union [Count of Units; unit: Fractures]
  None | 22 | 21 | 43
  Smoking | 5 | 4 | 9
  Obesity | 2 | 0 | 2
  Smoking and Obesity | 1 | 0 | 1
  Obesity and Leri-Weill Dischondrosteosis | 0 | 1 | 1
  Patient with paralized lower limbs following polio | 1 | 0 | 1
Fracture Cause [Count of Units; unit: Fractures]
  Domestic accident | 1 | 9 | 10
  Road traffic accident | 5 | 8 | 13
  Non-union | 11 | 3 | 14
  Domestic accident and Fall | 1 | 0 | 1
  Non-union and Pseudarthrosis after osteotomy in hip dysplasia | 2 | 0 | 2
  Fall | 4 | 0 | 4
  Trauma | 2 | 0 | 2
  Distorsion Trauma | 2 | 0 | 2
  Crush Trauma | 1 | 0 | 1
  New fracture on previous synthesis | 1 | 0 | 1
  Non-union and Nail breakage | 1 | 0 | 1
  Winter Sports accident | 0 | 5 | 5
  Correction following reduction and osteosynthesis performed at another center | 0 | 1 | 1
Open or Closed Fracture [Count of Units; unit: Fractures]
  Closed | 31 | 26 | 57
  Open | 0 | 0 | 0
Existence of Additional Fractures / Injuries [Count of Units; unit: Fractures]
  Yes | 4 | 0 | 4
  No | 27 | 26 | 53
AO/OTA Fracture Classification [Count of Units; unit: Fractures] — Each fracture = case was classified according to the AO/OTA Fracture Classification System. The system is a system introduced by the AO (Arbeitsgemeinschaft für Osteosynthesefragen) Foundation and the OTA (Orthopaedic Trauma Association) in order to assure a standardized and rational methodology of describing fractures and dislocations. It is an alphanumeric classification that can be applied throughout the skeleton, based on fracture location and morphology. Further information can be found: "https://ota.org/sites/files/2021-06/General%20A1%20Fracture%20Classifications.pdf"
  Fractures
    2U2A2 | 1 | 0 | 1
    4F2B1 | 2 | 0 | 2
    4F2B2 | 1 | 0 | 1
    12A1 | 1 | 0 | 1
    12A2 | 3 | 0 | 3
    12A3 | 3 | 0 | 3
    12B2 | 2 | 0 | 2
    12B3 | 1 | 0 | 1
    32A1 | 4 | 0 | 4
    32A2 | 3 | 0 | 3
    32A3 | 1 | 0 | 1
    32B2 | 1 | 0 | 1
    32B3 | 1 | 0 | 1
    32C2 | 1 | 0 | 1
    42A1 | 2 | 0 | 2
    42B1 | 1 | 0 | 1
    42B3 | 1 | 0 | 1
    87A2 | 2 | 0 | 2
    41A | 0 | 2 | 2
    41A1.2 | 0 | 1 | 1
    41A2 | 0 | 2 | 2
    41A3 | 0 | 1 | 1
    41A2.1 | 0 | 1 | 1
    41A2.2 | 0 | 7 | 7
    41A2.3 | 0 | 3 | 3
    41A3.2 | 0 | 1 | 1
    41A3.3 | 0 | 1 | 1
    41B1.1 | 0 | 2 | 2
    41B1.2 | 0 | 1 | 1
    41B2.1 | 0 | 1 | 1
    41B3.1 | 0 | 1 | 1
    41C1 | 0 | 1 | 1
    41C3.3 | 0 | 1 | 1
Operated Side [Count of Units; unit: Fractures]
  Left | 16 | 13 | 29
  Right | 15 | 13 | 28
Length of Hospital Stay [Mean (Standard Deviation); unit: days] | 4.3 (2.6) | 4.2 (2.2) | 4.2 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Performance: Fracture Healing
Description: Performance will be assessed by analyzing fracture healing radiographically or clinically. Timepoints at which the data will be collected will be summarized through means.
Time Frame: At last consultation visit either at minimum 6 months post-operative by radiographic assessment or, if no x-rays available, by clinical assessment at the follow-up phone call at minimum 1 year postoperative.
Measure: Count of Units; unit: Fractures
Units Other Than Participants: Fractures
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate
Number analyzed (Participants) | 30 | 26
Number analyzed (Fractures) | 31 | 26
Fractures
  Fracture healed | 29 | 26
  Fracture not healed | 2 | 0

2. Secondary Outcome: Product Safety (Number of Adverse Events, Serious Adverse Events, Adverse Device Effects and Serious Adverse Device Effects)
Description: Safety will be assessed by recording and analyzing the incidence and frequency of complications and adverse events. Timepoints at which the data will be collected will be summarized through means.
Time Frame: At operative evaluation, immediate post-operative evaluation, last consultation visit at minimum 6 months post-operative and at the follow-up phone call at minimum 1 year postoperative.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate: Adverse Events reported in 30 participants (31 cases) who meet the inclusion and none of the exclusion criteria and who received the Zimmer® Plates and Screws System in the Diaphysis.
- Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate: Adverse Events reported in 26 participants (26 cases) who meet the inclusion and none of the exclusion criteria and who received the Zimmer® Plates and Screws System in the Proximal Tibia.
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate
Number analyzed (Participants) | 31 | 26
Participants
  Adverse Events (AEs) | 0 | 3
  Serious Adverse Events (SAEs) | 0 | 3
  Adverse Device Effects (ADEs) | 0 | 0
  Serious Adverse Device Effects (SADEs) | 2 | 2
  No Adverse Events | 29 | 18

3. Secondary Outcome: Tegner Lysholm Knee Score (Proximal Tibia)
Description: Assessment of patient-reported outcome measures (PROMs):The Lysholm Knee Scoring Scale is an outcome measure addressing the following 8 symptoms; instability (25 points), pain (25 points), locking (15 points), swelling (10 points), stair climbing (10 points), limp (5 points), support (5 points), and squatting (5 points). Each of the 8 metrics uses different scoring systems. The total score is the sum of the 8 individual responses. Scores range from 0 (worse disability) to 100 (less disability).
Time Frame: Final follow-up visit at minimum 1 year postoperative.
Population: Patients implanted with the device in the Proximal Tibia.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate
Number analyzed (Participants) | 26
Score on a scale | 87.4 (19.0)

4. Secondary Outcome: Oxford Shoulder Score (OSS) (Proximal Humerus)
Description: Assessment of patient-reported outcome measures (PROMs): The Oxford Shoulder Score (OSS) is a patient-reported outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following TSA. The OSS consists of twelve questions covering function and pain associated with the shoulder. To calculate the total score, each question is scored from 5 (worst outcome) to 0 (best outcome) and the sum of all 12 items is reported with a maximum of 60, representing the worst score possible.
Time Frame: Final follow-up visit at minimum 1 year postoperative.
Population: No cases implanted with a Zimmer® Plates and Screws Proximal Humerus Plate were enrolled and analyzed in this study.
Groups:
- Patients Implanted With a Zimmer® Plates and Screws System Proximal Humerus Plate: 52 participants (52 cases) who meet the inclusion and none of the exclusion criteria and who received the Zimmer® Plates and Screws System in the Proximal Humerus.
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Proximal Humerus Plate
Number analyzed (Participants) | 0

5. Secondary Outcome: EuroQol Five-dimensional Health Questionnaire (EQ-5D-5L) (Diaphysis)
Description: Assessment of patient-reported outcome measures (PROMs): The EuroQol fivedimensional Health Questionnaire (EQ-5D) is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS), the highest score is 100 and the lowest score is 0. The questionnaire includes 5 questions referring to mobility, self-care, daily activities, pain/discomfort and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. In the derived EQ-5D-5L score, the highest score is 1 and the lowest score is -0.573.
Time Frame: Final follow-up visit at minimum 1 year postoperative.
Population: Patients implanted with the device in the Diaphysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate
Number analyzed (Participants) | 29
Score on a scale
  EQ-5D-5L Profile | 0.70 (0.30)
  Health State / VAS | 80.7 (20.9)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events from the date each subject was implanted up to 14.6 years after surgery, when the last follow-up was performed and patients completed the study.
Description: Adverse Events were collected in an Excel Spreadsheet, which gathered information of the date of occurrence, the nature of the adverse event, whether the device was involved, which treatment was used and the treatment outcome. No case was enrolled in the proximal humerus group and consequently no Adverse Events were reported in this group.
Arm/Group | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/30 | 5/26
Other Adverse Events (participants affected / at risk) | 0/30 | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate (N=30) | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate (N=26)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Development of pseudarthrosis after surgery with consequent reoperation with removal of fixation device and consequent new fixation.
Failure of device and new fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Bone fractured again at previous synthesis site, which required a revision surgery with consequent fracture healing.
Valgus knee deviation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Development of Valgus knee deviation after surgery, probably due to the localization of the fracture at the lateral hemiplate of the tibia. It required a distal femur varus osteotomy.
Infection (Infections and infestations) | 0 (0) | 2 (2) — Postoperative infections that had to be reoperated with removal of the devices.
New accident with a multifragmented fracture of the proximal tibia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Accident with a multifragmented fracture of the proximal tibia that required a reoperation with placement of a total knee prosthesis. The plate remained implanted, the proximal screws were removed.
Continued postoperative blood loss from the surgical wound (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Continuous postoperative blood loss from the surgical wound with consequent arteriography and embolization as treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With a Zimmer® Plates and Screws System Diaphysis Plate (N=30) | Patients Implanted With a Zimmer® Plates and Screws System Proximal Tibia Plate (N=26)
Postoperative anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Postoperative anemia that required treatment (iron supplementation/blood transfusion).

LIMITATIONS AND CAVEATS:
A limitation to this study is its retrospective design. Due to this, no patients implanted with a Zimmer® Plates and Screws System plate in the proximal humerus could be enrolled in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05215613/Prot_SAP_000.pdf